CLINICAL TRIAL: NCT00842764
Title: Minimally Invasive Holmium:YAG Laser Blepharoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Brian Wong, M.D., Ph.D., Professor Department of Otolaryngology, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20086593
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Lower Eyelid Entropion
Keywords: eyelid fat pads
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Holmium: YAG laser (Experimental): Subjects will go under minimally invasive Holmium: YAG laser blepharoplasty
  Interventions: Procedure: Holmium: YAG laser

INTERVENTIONS:
Procedure: Holmium: YAG laser — Minimally Invasive Holmium:YAG laser Blepharoplasty

SUMMARY:
The purpose of this research study is to is to evaluate the safety and effectiveness of the FDA approved Holmium:YAG laser for reducing lower eyelid bags.

DETAILED DESCRIPTION:
The researchers are interested in learning if the more precise Holmium:YAG laser can effectively tighten the orbital septum, a barrier of the orbit which holds fat in the bony orbit, while resulting in less unintentional surrounding damage and side effects.

ELIGIBILITY:
Inclusion Criteria:

* male/female 30 years and older
* have pronounced lower eyelid fat pads.

Exclusion Criteria:

* based on medical problems.
* Previous surgery or trauma to lower eyelid or orbit.
* pregnant or lactating.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Wong, M.D,PhD, Principal Investigator — Otolaryngology, UCIMC
Locations (1):
- UCIMC, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Holmium:YAG Laser: Subjects with minimally Invasive Holmium:YAG laser Blepharoplasty
Period: Overall Study
Arm/Group | Holmium:YAG Laser
Started | 7
Completed | 5
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Holmium:YAG Laser: Minimally Invasive Holmium:YAG laser Blepharoplasty
Arm/Group | Holmium:YAG Laser
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Lower Eyelid Bags.
Description: Preoperative and postoperative (postoperative visits were at day 1, 1 week, 1 month, and 2 months) .photographs were evaluated by 6 surgeons on a 5-point Likert scale which 1 indicates worsening, 2 means unchanged, 3 is mild improvement, 4 is moderate improvement, and 5 indicates complete correction.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Holmium:YAG Laser
Number analyzed (Participants) | 5
Participants
  Preoperative | 5
  Postoperative | 5

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Holmium:YAG Laser
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes